CLINICAL TRIAL: NCT01933399
Title: Comparison of Inextensible and Extensible Lumbosacral Orthoses for the Management of Episodes of Lower Back Pain
Brief Title: Comparison of Extensible and Inextensible Lumbosacral Orthoses for Lower Back Pain
Acronym: LSO LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, David Morrisette, Professor and Director, Division of Physical Therapy, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16527
Record Dates: First submitted 2013-06-24; First posted 2013-09-02 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Low Back Pain
Keywords: Low back pain; Back brace; Lumbar orthoses; Lumbosacral orthoses; Low back pain treatment
MeSH Terms: conditions — Low Back Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (Other): Medication based on physician prescriptions or overcounter use not germane to the study. Subjects also receive physical therapy for 2 weeks.
  Interventions: Other: Standard of Care
- Extensible lumbosacral orthoses plus standard of care (Experimental): This group receives a flexible/extensible lumbosacral orthosis, one that is commonly available over the counter
  Interventions: Other: Extensible LSO, a back support that is flexible
- Inextensible lumbosacral orthoses and standard of care (Experimental): This group receives an inextensible lumbosacral orthoses which leads to 14% increase in trunk stiffness compared to the other conditions.
  Interventions: Other: Inextensible LSO (stiff back support)

INTERVENTIONS:
Other: Inextensible LSO (stiff back support) — Cotton/nylon canvas back support with velcro fasteners.
  Arms: Inextensible lumbosacral orthoses and standard of care
Other: Extensible LSO, a back support that is flexible — Back support is constructed from lycra and neoprene with velcro fasteners.
  Arms: Extensible lumbosacral orthoses plus standard of care
Other: Standard of Care — Physician visit, physician advice, medications as determined by physician, over the counter medications, and physical therapy.
  Arms: Standard of Care

SUMMARY:
This study is designed to discern if the use of a lumbosacral orthesis (LSO, also call a back support) improves the short-term outcome of lower back pain. participants will receive standard care (physical therapy, physician treatment), with one group also receiving an extensible LSO, and another group receiving an inextensible LSO. The inextensible LSO has been shown to increase stiffness of the trunk in individuals while wearing it. The hypothesis is that the group wearing the inextensible LSO will have improved outcomes over the other two groups (standard care or standard care plus the extensible LSO).

ELIGIBILITY:
Inclusion Criteria:

* chief complaint of lower back pain, with or without lower extremity (LE) symptoms
* 150 subjects will be recruited from patients seeking treatment for lower back pain from spine specialty orthopaedic clinics, family practice physicians, and out-patient physical therapy clinics

Exclusion Criteria:

* Exclusion criteria are:
* previous spinal surgery
* workman's compensation or litigation is involved
* neurological disease or injury
* systemic inflammatory disease
* pulmonary disease which restricts breathing capacity
* current pregnancy
* acute fracture
* tumor or metastatic disease
* infection
* neurological disease
* the presence of pathological reflexes (e.g., Babinski)
* the presence of lower extremity pain upon cervical motion and / or the presence of two or more of the following signs of nerve compression: diminished lower extremity strength in a myotomal distribution, diminished sensation, and / or absence deep tendon reflexes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Morrisette, PT, PhD, Principal Investigator — Medical Unversity of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Extensible Lumbosacral Orthoses Plus Standard of Care | Inextensible Lumbosacral Orthoses and Standard of Care
Started | 29 | 32 | 37
Completed | 29 | 32 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Extensible Lumbosacral Orthoses Plus Standard of Care | Inextensible Lumbosacral Orthoses and Standard of Care | Total
Number analyzed (Participants) | 29 | 32 | 37 | 98
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 45.0 (16.6) | 48.8 (15.6) | 50.4 (14) | 48.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 20 | 60
  Male | 11 | 10 | 17 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 32 | 37 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 22 | 29 | 72
  White | 8 | 10 | 8 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 32 | 37 | 98

OUTCOME MEASURES:

1. Primary Outcome: Change Score in the Self-assessment of Disability as Measured by Oswestry Disability Index (ODI)
Description: Change score from baseline and the score at the second week. The Oswestry Disabilty Index is a 100 point self-assessment of disabilty due to lower back pain or complications from lower back pain. A score of 40 or more points is interpreted as signficant disability due to lower back pain. A score between 20 and 40 respresents disability, but the individual is still able to function to some degree with activities of daily living, but has to modify their behavior. A score less than 20 implies that the disabilty due to the lower back pain is not greatly impacting a wide range of functions. Compare score change to the minimal clinically important difference between the baseline and the 2nd week score, and the difference in the change scores across the 3 groups.
Time Frame: Baseline and 2 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard of Care | Extensible Lumbosacral Orthoses Plus Standard of Care | Inextensible Lumbosacral Orthoses and Standard of Care
Number analyzed (Participants) | 29 | 32 | 37
units on a scale | 2.4 [-2.2 to 7.1] | 8.1 [2.8 to 13.4] | 14.0 [8.2 to 19.8]
Statistical Analysis 1: Comparison: Standard of Care vs Inextensible Lumbosacral Orthoses and Standard of Care; ANCOVA Adjusted for baseline score; Test type: Superiority or Other; p = .01, ANCOVA; Mean Difference (Final Values) = 9.4, 95% CI 2-sided [2.2 to 16.6] — Difference in mean change in scores from baseline to follow-up by treatment group with no adjusment for baseline. a priori threshold determined to be .05. no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Standard of Care vs Extensible Lumbosacral Orthoses Plus Standard of Care; Test type: Superiority or Other; p = .16, ANCOVA — a priori threshold determined to be .05. no adjustments for multiple comparisons; Adjustment for baseline; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-2.0 to 12.6]

2. Secondary Outcome: Change Score in the Patient Specific Activity Scale
Description: Change score from baseline and the score at the second week. Compare score change to the minimal clinically important difference and analyze for statistical significance between the baseline and the 2nd week score, and the statistical difference in the change scores across the 3 groups. Scores from 0 to 10 with a higher score representing higher function and a lower score representing a decrease function.
Time Frame: Baseline and 2-weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard of Care | Extensible Lumbosacral Orthoses Plus Standard of Care | Inextensible Lumbosacral Orthoses and Standard of Care
Number analyzed (Participants) | 29 | 32 | 37
units on a scale | -0.4 [-1.3 to 0.4] | -1.2 [-1.9 to -0.5] | -1.8 [-2.6 to -1.0]
Statistical Analysis 1: Comparison: Standard of Care vs Inextensible Lumbosacral Orthoses and Standard of Care; Adjusted for baseline; Test type: Superiority or Other; p = 0.01, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.3 to -0.4]
Statistical Analysis 2: Comparison: Standard of Care vs Extensible Lumbosacral Orthoses Plus Standard of Care; Adjusted for baseline; Test type: Superiority or Other; p = .05, ANCOVA; Mean Difference (Final Values) = -1, 95% CI 2-sided [-2.1 to 0]

ADVERSE EVENTS:
Arm/Group | Standard of Care | Extensible Lumbosacral Orthoses Plus Standard of Care | Inextensible Lumbosacral Orthoses and Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32 | 0/37
Other Adverse Events (participants affected / at risk) | 0/29 | 0/32 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes